CLINICAL TRIAL: NCT04811313
Title: Impact of Tranexamic Acid Use on Blood Loss and Transfusion Rates After Hip Reconstruction in Children, A Randomized Controlled Trial
Brief Title: Tranexamic Acid in Pediatric Undergoing Proximal Femoral Osteotomies and/or Acetabular Osteotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abbas Hassan, lectrure of Anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: tranexamic acid in pediatric
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Intraoperative Blood Loss; Pediatric; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- T group (Active Comparator): each participant will receive 15 mg/kg of tranexamic acid diluted in a 10 mL syringe slowly over 10-15 minutes, 15 minutes before skin incision.
  Interventions: Drug: Tranexamic acid
- TC group (Active Comparator): each participant will receive 10 mg/kg of tranexamic acid diluted in a 5 mL syringe slowly over 5 minutes, 15 minutes before skin incision, and A caudal epidural block with 1 mL/kg of 0.25% bupivacaine.
  Interventions: Drug: Tranexamic acid; Procedure: caudal epidural block
- C group (Active Comparator): each participant will receive a caudal epidural block with 1 mL/kg of 0.25% bupivacaine.
  Interventions: Procedure: caudal epidural block
- P group (Placebo Comparator): participants will receive the regular standard care without adding tranexamic acid or caudal epidural block
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — patients treated with TXA will have reduced blood loss and transfusion requirements compared with those who did not receive TXA
  Other Names: Kapron
  Arms: T group; TC group
Procedure: caudal epidural block — regional anesthesia in orthopedic procedures are known to help reduction of intraoperative blood loss
  Other Names: bupivacaine 0.25%
  Arms: C group; TC group
Other: Placebo — participants will receive standard care but neither TXA nor caudal epidural block
  Arms: P group

SUMMARY:
Surgical hip reconstruction reduces the hip joint through soft tissue releases and osteotomies of the femur and/or pelvis. Blood loss and subsequent blood transfusion are normal consequences of hip reconstruction.

DETAILED DESCRIPTION:
the use of antifibrinolytics (AFs) to limit blood loss peri-operatively has been popularized in certain subspecialties. AFs have been studied extensively in adults undergoing various orthopedic procedures including spine and total joint arthroplasty, and have been proven to reduce blood loss and reduce the risk of blood transfusion. Similarly, AFs are used in pediatric patients undergoing cardiac surgery as well as craniofacial operations. Tranexamic acid (TXA) is a synthetic anti-fibrinolytic agent that works by reversibly blocking plasminogen and thereby promoting hemostasis through the prevention of fibrin degradation. Current literature investigating the safety and effectiveness of TXA in children undergoing orthopedic procedures is limited.

We hypothesize that patients treated with TXA will have reduced blood loss and transfusion requirements compared with those who did not receive TXA.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II
* Scheduled for acetabular osteotomy and/or proximal femoral derotation osteotomies.

Exclusion Criteria:

* Patient's guardian refusal to participate in the study.
* Children known to have pre-existing bleeding or coagulation disorders.
* Children with anemia; defined according to (WHO ) cutoffs as Hb level<11g/dl for girls and <12g/dl for boys
* History of epilepsy.
* History of renal insufficiency or failure

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
amount of intraoperative blood loss | 24 hours
  calculated from the fall in red blood cell volume

SECONDARY OUTCOMES:
Rate of blood transfusion | 24 hours
  either intraoperative or postoperative blood transfusion
Incidence of adverse effects or complications of TXA | 24 hours
  e.g. thromboembolic events or perioperative seizures will be managed and recorded
length of hospital stay | 24 hours
  readiness for hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Sleem, M.D., Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt